CLINICAL TRIAL: NCT03263247
Title: Randomized Double Blind Study on the Efficacy of Cognitive Training in Patients With Mild Cognitive Impairment Using fMRI.
Brief Title: Cognitive Training in Patients With MCI Using fMRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: São Paulo State University (Other)
Collaborators: Ricardo Nitrini (Unknown); Sonia Brucki (Unknown); Maira Okada de Oliveira (Unknown); Edson Amaro Junior (Unknown); Maria da Graca M Martin (Unknown); Rodolfo dos Anjos (Unknown); Camila Carneiro Pedroza (Unknown); Ana Carolina Cruz (Unknown); Aline Gisele Gonçalves (Unknown); Leticia Nery Celino de Souza Pak (Unknown); Letícia Ferreira da Mota (Unknown); Paulo Rodrigo Bazán (Unknown); Isabella Maria Bello Avolio (Unknown)
Responsible Party: Principal Investigator, Eliane Mioto, Prof. Dr Eliane C Miotto, São Paulo State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MCI cognitive training
Record Dates: First submitted 2017-08-24; First posted 2017-08-28 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Visual Imaging Training (Experimental): Participants will receive visual imaging training to facilitate learning of written information.
  Intervention: Visual Imaging Training in individual sessions
  Interventions: Behavioral: Memory Training
- Psychoeducation (Active Comparator): Participants will receive information about memory functioning and aging.
  Intervention: behavioral: Psychoeducation in individual sessions
  Interventions: Behavioral: Psychoeducation
- Alphabet Search (Experimental): Participants will receive alphabet search training.
  Intervention: Alphabet Search in individual sessions
  Interventions: Behavioral: Alphabet search

INTERVENTIONS:
Behavioral: Memory Training
  Arms: Visual Imaging Training
Behavioral: Psychoeducation
  Arms: Psychoeducation
Behavioral: Alphabet search
  Arms: Alphabet Search

SUMMARY:
The current project aims to investigate the efficacy of the visual imaging training (VIT) and alphabet search training in comparison to an active control intervention, namely psychoeducation information (PI) using fMRI in patients with amnestic mild cognitive impairment (MCI) and healthy elderly controls (HE). MCI patients will be grouped according to biomarkers (PET PIB, PET FDG and liquor).

DETAILED DESCRIPTION:
We will include 30 subjects with amnestic mild cognitive impairment (MCI) single domain or multiple domain clinical diagnostic, over 60 years old, recruited through the Cognitive and Behavioral Neurology Group ambulatory of University of Sao Paulo General Hospital. We will also include 30 healthy subjects, over 60 years old, recruited in the community. All the participants will be evaluated by neurologists specialized in cognitive neurology and subjected to a neuropsychological assessment. The 30 participants with MCI and 30 healthy subjects will be divided in 6 groups: the G1 MCI group (N=10) will receive 4 sessions of visual imaging training; the G2 control group (N=10) will receive 4 sessions of visual imaging training; the G3 MCI group (N=10) will receive psychoeducation intervention; the G4 control group (N=20) will receive psychoeducation intervention; the G5 MCI group (N=10) will receive cognitive training with alphabet search training and the G6 control group will receive cognitive training with alphabet search training. This will be a longitudinal, randomized, double blind study. MCI patients will be grouped according to biomarkers (PET PIB, PET FDG and liquor).

ELIGIBILITY:
Inclusion Criteria:

* Portuguese as native and preferred language; A minimum of 4 years of education; MRI-compatible; Right-handed individuals; Normal corrected vision and hearing; Estimated intelligence average or above (≥ 80 IQ); Amnestic Mild Cognitive Impairment identified by a doctor and neuropsychological tests; Able to give informed consent.

Exclusion Criteria:

* History of neurological disorder; History of serious systemic disease; History of severe mental illness; Current untreated alcohol or substance abuse; Medical conditions that compromise in any way the central nervous system; Presence of visual impairment and / or hearing to preclude cognitive testing; Presence of contraindications to MRI exam; Findings in structural MRI that can interfere with the results of the study

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-01-02 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in functional magnetic resonance imaging (fMRI) | Baseline and after 4 weeks of intervention fMRI correlates of behavioral performance
  fMRI correlates of behavioral performance
Changes in memory and language measures | Baseline and after 4 weeks of intervention - generalization
  Improvement in Logical Memory Test I and II results and naming tests

SECONDARY OUTCOMES:
Changes in perception of memory performance | Baseline, within four weeks after intervention
  Multifactorial Memory Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil